CLINICAL TRIAL: NCT06116318
Title: Absolute Quantification of c-Kit Mutation as MRD in Acute Myeloid Leukemia: a Prospective Observational Study
Brief Title: A Study of c-Kit Mutation as MRD in Acute Myeloid Leukemia
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QT2023009
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: C-KIT Mutation
Keywords: Acute myeloid leukemia; c-Kit mutation; MRD
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- MRD negative: c-Kit mutation tested negative
- MRD L1: MRD detection at low level-1：<0.001%
- MRD L2: MRD detection at low level-2：0.001%≤c-Kit MRD<0.01%
- MRD L3: detection at low level-3：0.01%≤c-Kit MRD<0.1%
- MRD positive: MRD positive：c-Kit MRD≥0.1%

SUMMARY:
C-Kit is involved in an essential pathway of disease occurrence and is closely related to the poor prognosis of patients. However, the clinical significance of c-Kit mutation as molecular MRD monitoring is still unclear. What are the differences and advantages of using c-Kit mutation as MRD in prognostic assessment compared with other MRDs (MFC or RUNX1::RUNX1T1) widely used today? Existing data suggest that patients with one positive and one negative MRD results obtained by two different techniques have a higher risk of recurrence than patients with two negative MRD results but a lower risk of recurrence than patients with two positive MRD results. Therefore, can combining multiple MRD markers, including c-Kit mutations, overcome the shortcomings of a single molecular marker as MRD monitoring? Therefore, this project intends to confirm the clinical significance of quantitative detection of c-Kit mutation as MRD in acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the diagnostic criteria(WHO 2016 criteria) of AML and have c-Kit D816 mutation. And receive treatment.

Exclusion Criteria:

Patients with other factors which were considered unsuitable to participate in the study by the investigators

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute myeloid leukemia confirmed by bone marrow cell morphology, immunology, and genetics. And c-Kit D816 mutation was positive.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
CIR | Within 5 years after treatment
  cumulative incidence of recurrence

SECONDARY OUTCOMES:
OS | Within 5 years after treatment
  Overall Survival Rate
RFS | Within 5 years after treatment
  Relapse-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China